CLINICAL TRIAL: NCT02724800
Title: Implementation of Brief Insomnia Treatments - Clinical Trial
Acronym: iBIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Adam Bramoweth, Research Health Scientist, VA Pittsburgh Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00001553; 1IK2HX001548-01A2 (NIH)
Record Dates: First submitted 2016-03-21; First posted 2016-03-31 (Estimated); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Chronic Insomnia
Keywords: Insomnia; Veterans; Cognitive Behavioral Therapy for Insomnia; Brief Behavioral Treatment for Insomnia; Comparative Effectiveness Research
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBTI (Active Comparator): CBTI consists of five in-person sessions within an eight week period. Topics covered include: sleep education, stimulus control, sleep restriction, relaxation strategies, cognitive therapy, and sleep hygiene.
  Interventions: Behavioral: CBTI
- BBTI (Active Comparator): BBTI consists of one in-person session with three weekly follow-up sessions (in-person or phone) in a four week period. Topics covered include: sleep education, stimulus control, and sleep restriction.
  Interventions: Behavioral: BBTI

INTERVENTIONS:
Behavioral: CBTI — 28 Veterans with chronic insomnia will be randomized to CBTI. The intervention will be delivered in 5 face-to-face session within an 8 week time period. The intervention will be delivered at the VA Pittsburgh Healthcare System. Treatment visits will last approximately 45 minutes.
  Other Names: Cognitive Behavioral Therapy for Insomnia
  Arms: CBTI
Behavioral: BBTI — 28 Veterans with chronic insomnia will be randomized to BBTI. The intervention will be delivered over 4 consecutive weeks, which include individual face-to-face visits on Weeks 1 and 3 (option for telephone), and telephone appointments on Weeks 2 and 4. Interventions will be delivered at the VA Pittsburgh Healthcare System. The duration of the first treatment visit is approximately 45-minutes, and the follow-up visit on Week 3 will last no more than 30 minutes. Brief (<20 minutes) telephone sessions will be conducted on Weeks 2 and 4.
  Other Names: Brief Behavioral Treatment for Insomnia
  Arms: BBTI

SUMMARY:
The purpose of this study is to directly compare the effectiveness of two interventions for insomnia: Brief Behavioral Treatment for Insomnia (BBTI) vs. Cognitive Behavioral Therapy for Insomnia (CBTI).

DETAILED DESCRIPTION:
Cognitive Behavioral Therapy for Insomnia (CBTI) is the evidence-based first line treatment for chronic insomnia. Randomized controlled trials and meta-analyses have established that CBTI is efficacious and effective. Despite the strong evidence for CBTI, chronic insomnia remains under-treated among Veterans because of several barriers that limit access to behavioral treatments. In recent years, the VA has taken substantial measures to train more clinicians to provide insomnia treatment; however, a deficit in treatment availability remains. In 2011, the VA began to train clinicians in CBTI as part of the VA's Evidence Based Psychotherapy (EBP) training program, with a goal to train 1000 clinicians. Even with 1000 VA clinicians trained in CBTI, a shortage of clinicians will likely remain due to the high prevalence of insomnia. High prevalence and a shortage of clinicians prevent the VA from meeting the care demand of Veterans with insomnia. While the CBTI roll-out is a significant investment from the VA, additional mechanisms, such as dissemination and implementation of other evidence-based treatments for insomnia with fewer implementation barriers, must be considered to address the high prevalence of insomnia.

The in-person delivery and length of treatment for CBTI may be one of barriers to accessing care. Briefer protocols that use multiple delivery modalities have recently been developed and may help to increase session attendance and treatment completion. These shorter insomnia treatments are often referred to as Brief Behavioral Treatment for Insomnia (BBTI) and consist of ≤4 sessions. Besides fewer and briefer sessions, and utilizing both in-person and phone delivery of treatment, BBTI also emphasizes the behavioral components of CBTI (i.e., stimulus control and sleep restriction) rather than a combined approach focusing on both behavioral and cognitive components. BBTI is efficacious in adults-studies with older adults and Veterans found BBTI resulted in a significant decrease in insomnia severity with Cohen's d effect sizes in the moderate to large range. Like CBTI, BBTI significantly improves insomnia severity and may also help to improve secondary outcomes like depression and anxiety.

Integration of newer insomnia treatments, like BBTI, will first depend on establishing its evidence directly compared to CBTI. Effectiveness trials of BBTI, especially those conducted with military Veterans in typical VA settings, have yet to be conducted. Before BBTI can be broadly implemented and integrated into the VA, it needs to be established as a clinically effective treatment for insomnia among Veterans and a statistically non-inferior treatment (not necessarily better or worse) for Veterans compared to CBTI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old and older
2. Military Veteran
3. Insomnia Severity Index (ISI) ≥15 & Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for insomnia disorder
4. If using sleep medications, medication and dosage have not been changed in the past month, and will remain unchanged for the duration of the treatment phase of the study (i.e., 4-8 weeks)
5. If using other psychotropic medications, medication and dosage have not been changed in the past 2 months, and will remain unchanged for the duration of the treatment phase of the study (i.e., 4-8 weeks)

Exclusion Criteria:

1. Untreated, current, and severe PTSD as determined by the Structured Clinical Interview for DSM-5 (SCID)
2. Untreated, current, and severe Major Depressive Disorder as determined by the SCID
3. Current/Past Psychotic or Bipolar disorder
4. Current substance or alcohol use disorder as determined by the SCID
5. Current unstable medical condition
6. Hospitalization in the previous 1 month for a medical condition or surgery for which recovery overlaps with the study onset and duration
7. Seizure disorder, open skull brain injury, or moderate to severe traumatic brain injury (TBI)
8. Current, untreated, sleep disorders such as nightmare disorder, restless legs syndrome, circadian rhythm disorder (or shift work), or a suspected sleep disorder requiring polysomnographic assessment, such as obstructive sleep apnea or periodic leg movements as determined by the South Texas Research Organizational Network Guiding Studies on Trauma and Resilience (STRONG STAR) Clinical Interview for DSM-5 Sleep-Wake Disorders and/or the STOP-BANG questionnaire
9. Moderate to severe cognitive impairment (St. Louis University Mental Status [SLUMS] exam ≤20) and/or diagnosis in medical record indicative of moderate to severe cognitive impairment
10. Unstable environment that is not in one's control (e.g., homeless, temporary group home, care taking duties at night)
11. Pregnancy and/or breast-feeding

STOP-BANG is not a true acronym but indicates the symptoms each item assess:

* S-snores T-tired/sleepy O-observed apneas P-high blood pressure
* B-body mass index A-age N-neck circumference G-gender

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Bramoweth AD, Lederer LG, Youk AO, Germain A, Chinman MJ. Brief Behavioral Treatment for Insomnia vs. Cognitive Behavioral Therapy for Insomnia: Results of a Randomized Noninferiority Clinical Trial Among Veterans. Behav Ther. 2020 Jul;51(4):535-547. doi: 10.1016/j.beth.2020.02.002. Epub 2020 Feb 20. PMID 32586428
- [Derived] Bramoweth AD, Germain A, Youk AO, Rodriguez KL, Chinman MJ. A hybrid type I trial to increase Veterans' access to insomnia care: study protocol for a randomized controlled trial. Trials. 2018 Jan 26;19(1):73. doi: 10.1186/s13063-017-2437-y. PMID 29373993

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 92 participants met initial eligibility criteria and signed informed consent to participate in the study.
  However, only 63 participants met full criteria to participate and were randomized to a treatment arm.
Groups:
- Cognitive Behavioral Therapy for Insomnia (CBTI): Cognitive Behavioral Therapy for Insomnia (CBTI) consisted of five in-person sessions within an eight week period. Topics covered included: sleep education, stimulus control, sleep restriction, relaxation strategies, cognitive therapy, and sleep hygiene.
  CBTI: 32 Veterans with chronic insomnia were randomized to CBTI. The intervention was delivered in 5 face-to-face session within an 8 week time period. The intervention was delivered at the VA Pittsburgh Healthcare System. Treatment visits lasted approximately 45 minutes.
- Brief Behavioral Treatment for Insomnia (BBTI): Brief Behavioral Treatment for Insomnia (BBTI) consisted of one in-person session with three weekly follow-up sessions (in-person or phone) in a four week period. Topics covered included: sleep education, stimulus control, and sleep restriction.
  BBTI: 31 Veterans with chronic insomnia were randomized to BBTI. The intervention was delivered within 5 weeks, which included individual face-to-face visits on Weeks 1 and 3 (option for telephone) and telephone appointments on Weeks 2 and 4. The intervention was delivered at the VA Pittsburgh Healthcare System. The duration of the first treatment visit was approximately 45-minutes, and the follow-up visit on Week 3 was approximately 30 minutes. Brief (<20 minutes) telephone sessions were conducted on Weeks 2 and 4.
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy for Insomnia (CBTI) | Brief Behavioral Treatment for Insomnia (BBTI)
Started | 32 | 31
Completed | 15 | 22
Not Completed | 17 | 9

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Cognitive Behavioral Therapy for Insomnia (CBTI): CBTI consisted of five in-person sessions within an eight week period. Topics covered included: sleep education, stimulus control, sleep restriction, relaxation strategies, cognitive therapy, and sleep hygiene.
  CBTI: 32 Veterans with chronic insomnia were randomized to CBTI. The intervention was delivered in 5 face-to-face session within an 8 week time period. The intervention was delivered at the VA Pittsburgh Healthcare System. Treatment visits lasted approximately 45 minutes.
- Brief Behavioral Treatment for Insomnia (BBTI): BBTI consisted of one in-person session with three weekly follow-up sessions (in-person or phone) in a four week period. Topics covered included: sleep education, stimulus control, and sleep restriction.
  BBTI: 31 Veterans with chronic insomnia were randomized to BBTI. The intervention was delivered within 5 weeks, which included individual face-to-face visits on Weeks 1 and 3 (option for telephone) and telephone appointments on Weeks 2 and 4. The intervention was delivered at the VA Pittsburgh Healthcare System. The duration of the first treatment visit was approximately 45-minutes, and the follow-up visit on Week 3 was approximately 30 minutes. Brief (<20 minutes) telephone sessions were conducted on Weeks 2 and 4.
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy for Insomnia (CBTI) | Brief Behavioral Treatment for Insomnia (BBTI) | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (15.2) | 56.8 (13.7) | 55.1 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 28 | 29 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 26 | 24 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 31 | 63
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: score on a scale] — Insomnia Severity Index (ISI) 0-28; 0-7 (no symptoms), 8-14 (sub-threshold symptoms), 15-21 (moderately severe), 22-28 (severe) high scores indicate worse outcome/greater severity
  score on a scale | 20.6 (3.7) | 19.8 (3.5) | 20.22 (3.59)
Pittsburgh Sleep Quality Index (PSQI) [Mean (Standard Deviation); unit: score on a scale] — Pittsburgh Sleep Quality Index (PSQI) 0-21 higher score indicates worse sleep quality, >5 indicates poor quality sleep
  score on a scale | 12.9 (3.5) | 12.3 (4.0) | 12.6 (3.7)
Patient Global Impression of Change (PGIC) [Mean (Standard Deviation); unit: score on a scale] — Patient Global Impression of Change (PGIC) 1-7 higher score indicative of greater subjective improvement
  score on a scale | 1.9 (1.3) | 1.7 (1.1) | 1.8 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index (ISI)
Description: Insomnia Severity Index (ISI) 0-28; 0-7 (no symptoms), 8-14 (sub-threshold symptoms), 15-21 (moderately severe), 22-28 (severe) high scores indicate worse outcome/greater severity
Time Frame: post-treatment (BBTI: week 5; CBTI: week 6-9)
Population: Participants who completed post-treatment ISI
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CBTI: CBTI consisted of five in-person sessions within an eight week period. Topics covered included: sleep education, stimulus control, sleep restriction, relaxation strategies, cognitive therapy, and sleep hygiene.
  CBTI: 32 Veterans with chronic insomnia were randomized to CBTI. The intervention was delivered in 5 face-to-face session within an 8 week time period. The intervention was delivered at the VA Pittsburgh Healthcare System. Treatment visits lasted approximately 45 minutes.
- BBTI: BBTI consisted of one in-person session with three weekly follow-up sessions (in-person or phone) in a four week period. Topics covered included: sleep education, stimulus control, and sleep restriction.
  BBTI: 31 Veterans with chronic insomnia were randomized to BBTI. The intervention was delivered within 5 weeks, which included individual face-to-face visits on Weeks 1 and 3 (option for telephone) and telephone appointments on Weeks 2 and 4. The intervention was delivered at the VA Pittsburgh Healthcare System. The duration of the first treatment visit was approximately 45-minutes, and the follow-up visit on Week 3 was approximately 30 minutes. Brief (<20 minutes) telephone sessions were conducted on Weeks 2 and 4.
Arm/Group | CBTI | BBTI
Number analyzed (Participants) | 17 | 22
score on a scale | 9.6 (4.9) | 11.0 (6.5)
Statistical Analysis 1: Comparison: CBTI vs BBTI; Test type: Non-Inferiority — non-inferiority margin = 3.43; p < 0.05, Mixed Models Analysis — a priori; Mean Difference (Net) = 2.2, 95% CI 2-sided [-0.9 to 5.6]

2. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: Patient Health Questionnaire (PHQ-9) 0-27; 0-5 (minimal), 6-10 (mild), 11-15 (moderate), 16-20 (moderate-severe), 21-27 (severe) high scores indicate worse outcome/greater severity
Time Frame: post-treatment (BBTI: week 5; CBTI: week 6-9)
Population: Participants who completed post-treatment PHQ-9 (no sleep item)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBTI | BBTI
Number analyzed (Participants) | 17 | 22
score on a scale | 5.1 (4.3) | 5.1 (4.9)

3. Secondary Outcome: Generalized Anxiety Disorder (GAD-7)
Description: Generalized Anxiety Disorder (GAD-7) 0-21; 0-5 (minimal), 6-10 (mild), 11-15 (moderate), 16-21 (severe) high scores indicate worse outcome/greater severity
Time Frame: post-treatment (BBTI: week 5; CBTI: week 6-9)
Population: Participants who completed post-treatment GAD-7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBTI | BBTI
Number analyzed (Participants) | 17 | 22
score on a scale | 5.2 (3.5) | 5.0 (4.7)

4. Secondary Outcome: PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (PCL-5)
Description: PTSD Checklist for DSM-5 (PCL-5) 0-76 (sleep item removed), higher scores indicate greater PTSD severity >33, likely PTSD diagnosis
Time Frame: post-treatment (BBTI: week 5; CBTI: week 6-9)
Population: Participants who completed post-treatment PCL-5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBTI | BBTI
Number analyzed (Participants) | 17 | 22
score on a scale | 14.2 (14.1) | 14.8 (13.4)

5. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Scale
Description: PROMIS Fatigue Scale 33.4 - 76.8 (T-score) The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a participant with a T-score of 50 is equal to the mean and a T-score of 40 is one SD below the mean. Scores less than 50 indicate less fatigue symptoms than an age and gender matched healthy population and scores greater than 50 indicate greater fatigue symptoms than an age and gender matched healthy population.
Time Frame: post-treatment (BBTI: week 5; CBTI: week 6-9)
Population: Participants who completed post-treatment PROMIS Fatigue
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | CBTI | BBTI
Number analyzed (Participants) | 17 | 22
T-score | 53.4 (9.3) | 54.2 (11.4)

6. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health
Description: PROMIS Global Health Physical Health: 16.2 - 67.7 (T-score) Mental Health: 21.2 - 67.6 (T-score) The T-score re-scales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a participant with a T-score of 50 is equal to the mean and a T-score of 40 is one SD below the mean. Scores less than 50 indicate worse quality of life than an age and gender matched healthy population and scores greater than 50 indicate better quality of life than an age and gender matched healthy population.
Time Frame: post-treatment (BBTI: week 5; CBTI: week 6-9)
Population: Participants who completed post-treatment PROMIS Global Health
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | CBTI | BBTI
Number analyzed (Participants) | 17 | 22
T-score
  Physical Health (post-tx) | 41.8 (8.3) | 41.4 (8.1)
  Mental Health (post-tx) | 45.6 (8.6) | 45.8 (9.2)

7. Secondary Outcome: Work and Social Adjustment Scale (WSAS)
Description: Work and Social Adjustment Scale (WSAS) 0-40 higher scores indicate worse functioning
Time Frame: post-treatment (BBTI: week 5; CBTI: week 6-9)
Population: Participants who completed post-treatment WSAS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBTI | BBTI
Number analyzed (Participants) | 17 | 22
score on a scale | 10.8 (9.1) | 12.5 (10.1)

8. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: Pittsburgh Sleep Quality Index (PSQI) 0-21 higher score indicates worse sleep quality, >5 indicates poor quality sleep
Time Frame: post-treatment (BBTI: week 5; CBTI: week 6-9)
Population: Participants that completed post-treatment PSQI assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBTI | BBTI
Number analyzed (Participants) | 17 | 22
score on a scale | 6.8 (3.5) | 8.4 (4.3)
Statistical Analysis 1: Comparison: CBTI vs BBTI; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 2.3

9. Secondary Outcome: Epworth Sleepiness Scale (ESS)
Description: Epworth Sleepiness Scale (ESS) 0-24 higher score indicates greater sleepiness, >10 indicates excessive daytime sleepiness
Time Frame: post-treatment (BBTI: week 5; CBTI: week 6-9)
Population: Participants who completed post-treatment ESS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBTI | BBTI
Number analyzed (Participants) | 17 | 22
score on a scale | 9.2 (4.7) | 9.4 (5.0)

10. Secondary Outcome: Dysfunctional Beliefs and Attitudes About Sleep (DBAS)
Description: Dysfunctional Beliefs and Attitudes About Sleep (DBAS) 0-160 reported as mean score (sum of items answered / 10 for a range 0-16) higher scores indicate greater dysfunctional beliefs and attitudes
Time Frame: post-treatment (BBTI: week 5; CBTI: week 6-9)
Population: Participants who completed post-treatment DBAS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBTI | BBTI
Number analyzed (Participants) | 17 | 22
score on a scale | 4.6 (1.9) | 4.4 (1.6)

11. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: Patient Global Impression of Change (PGIC) 1-7 higher score indicative of greater subjective improvement
Time Frame: post-treatment (BBTI: week 5; CBTI: week 6-9)
Population: Participants that completed post-treatment PGIC
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBTI | BBTI
Number analyzed (Participants) | 17 | 22
score on a scale | 5.0 (1.6) | 4.7 (1.9)
Statistical Analysis 1: Comparison: CBTI vs BBTI; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 0.3

12. Secondary Outcome: Sleep Diary
Description: The Sleep Diary measures common sleep variables important for tracking and changing sleep behaviors Sleep Onset Latency (SOL) - lower is better Wake After Sleep Onset (WASO) - lower is better Early Morning Awakenings (EMA) - lower is better Total Wake Time (TWT) - lower is better Total Sleep Time (TST) - higher is better Time in Bed (TIB) - value depends on TWT and TST
Time Frame: post-treatment (BBTI: week 5; CBTI: week 6-9)
Population: Participants who completed post-treatment Sleep Diaries
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | CBTI | BBTI
Number analyzed (Participants) | 12 | 9
minutes
  Sleep Onset Latency (SOL) | 23.5 (22.0) | 20.8 (10.9)
  Wake After Sleep Onset (WASO) | 27.4 (33.0) | 18.5 (15.9)
  Early Morning Awakenings (EMA) | 10.7 (14.7) | 12.8 (20.2)
  Total Wake Time (TWT) | 78.9 (35.2) | 67.5 (29.9)
  Total Sleep Time (TST) | 410.3 (67.6) | 381.6 (60.0)
  Time in Bed (TIB) | 489.3 (77.7) | 449.0 (37.6)

13. Secondary Outcome: Sleep Diary - Sleep Efficiency
Description: The Sleep Diary measures common sleep variables important for tracking and changing sleep behaviors Sleep Efficiency (total sleep time [TST] / time in bed [TIB]) x 100 - higher is better
Time Frame: post-treatment (BBTI: week 5; CBTI: week 6-9)
Population: Participants who completed post-treatment Sleep Diaries
Measure: Mean (Standard Deviation); unit: percentage of TST / TIB
Arm/Group | CBTI | BBTI
Number analyzed (Participants) | 12 | 9
percentage of TST / TIB | 83.9 (6.1) | 84.6 (7.8)

14. Secondary Outcome: Sleep Diary - Sleep Quality
Description: The Sleep Diary measures common sleep variables important for tracking and changing sleep behaviors Sleep Quality (SQ) 1-5 higher is better
Time Frame: post-treatment (BBTI: week 5; CBTI: week 6-9)
Population: Participants who completed post-treatment Sleep Diaries
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBTI | BBTI
Number analyzed (Participants) | 12 | 9
score on a scale | 3.4 (0.7) | 2.8 (0.5)

ADVERSE EVENTS:
Time Frame: baseline to 12-month follow-up (approximately 57-60 weeks)
Arm/Group | CBTI | BBTI
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31

LIMITATIONS AND CAVEATS:
In general, higher than expected dropout leading to smaller number of participants analyzed.

For sleep diaries, higher than expected dropout and poor completion at post-treatment resulted in small number analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/00/NCT02724800/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/00/NCT02724800/Prot_SAP_001.pdf